CLINICAL TRIAL: NCT02627053
Title: Treatment of Portal, Mesenteric, and Splenic Vein Thrombosis With Rivaroxaban. A Pilot, Prospective Cohort Study
Brief Title: Treatment of Splanchnic Vein Thrombosis With Rivaroxaban. A Pilot, Prospective Cohort Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Walter Ageno, Associate Professor of Medicine, Università degli Studi dell'Insubria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIVASVT-100
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Portal Vein Thrombosis; Mesenteric Vein Thrombosis; Splenic Vein Thrombosis
MeSH Terms: conditions — Mesenteric Ischemia | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rivaroxaban (Experimental)
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: rivaroxaban

SUMMARY:
Anticoagulant therapy is generally recommended for all patients presenting with acute symptomatic splanchnic vein thrombosis, starting with either low-molecular weight heparin (LMWH) or unfractionated heparin and continuing with the vitamin K antagonists in most patients. Rivaroxaban is approved for the treatment of deep vein thrombosis and pulmonary embolism, but no studies have assessed the safety of rivaroxaban in the setting of splanchnic vein thrombosis. The investigators aim to collect prospective information on the safety of rivaroxaban in a pilot cohort of 100 patients with acute splanchnic vein thrombosis without liver cirrhosis.

DETAILED DESCRIPTION:
Patients with splanchnic vein thrombosis are at increased risk of recurrent VTE and bleeding. Routine anticoagulation with unfractionated heparin or low molecular weight heparin followed by warfarin is recommended in this setting, but limited data is available to support this recommendation and more than 20% of these patients do not receive antithrombotic treatment due the fear for bleeding complications. The pharmacokinetic and pharmacodynamic characteristics of rivaroxaban make this drug an ideal alternative therapeutic strategy for the treatment of patients with SVT. Thanks to the oral route of administration, the short half-life, the high bioavailability, the predictable dose-response and the lack of effects on platelet activity, rivaroxaban could result as an important alternative to both LMWH and warfarin in the acute and long-term treatment of SVT patients. Furthermore, the analysis of phase III studies conducted in patients with DVT or PE have shown a better safety profile of rivaroxaban as compared to standard of treatment. This observed benefit in the safety profile of rivaroxaban would be extremely relevant in the treatment of patients with SVT. In this prospective cohort study, patients presenting with acute SVT will receive rivaroxaban 15 mg bid for 3 weeks followed by rivaroxaban 20 mg od for a total of 3 months. The primary safety and efficacy outcomes will be measured at 3 months.

ELIGIBILITY:
Inclusion criteria:

* Consecutive patients aged 18 years or older
* first episode of symptomatic, objectively diagnosed PVT, MVT, or spVT
* signed informed consent.

Exclusion criteria:

* known liver cirrhosis (biopsy proven or with clinical, laboratory, or imaging evidence of chronic liver disease, within a context of chronic alcoholism, viral hepatitis, autoimmunity, Wilson's disease, iron overload)
* alanine aminotransferase level that is three times the upper limit of the normal range or higher
* Budd-Chiari syndrome
* previous or ongoing vatical bleeding
* presence of portal vein cavernoma at the time of diagnosis
* anticipated abdominal surgical procedure
* known bleeding diathesis
* platelet count <100.000 mm3
* creatinine clearance <30 mL/min (Cockroft-Gault formula)
* life expectancy of less than 3 months
* expected inability to take oral medications
* concomitant treatment with azole antimycotics and human immunodeficiency virus protease inhibitors - treatment with therapeutic doses of LMWH or UFH for more than 7 days
* ongoing treatment with VKA
* pregnancy or lactation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Major bleeding | 3 months

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (3):
  - McMaster University, Hamilton
  - University of Western Ontario, London
  - University of Ottawa, Ottawa
- Ospedale di Circolo, Varese, Italy

REFERENCES:
- [Derived] Ageno W, Beyer Westendorf J, Contino L, Bucherini E, Sartori MT, Senzolo M, Grandone E, Santoro R, Carrier M, Delluc A, De Stefano V, Pomero F, Donadini MP, Tosetto A, Becattini C, Martinelli I, Nardo B, Bertoletti L, Di Nisio M, Lazo-Langner A, Schenone A, Riva N. Rivaroxaban for the treatment of noncirrhotic splanchnic vein thrombosis: an interventional prospective cohort study. Blood Adv. 2022 Jun 28;6(12):3569-3578. doi: 10.1182/bloodadvances.2022007397. PMID 35439303